CLINICAL TRIAL: NCT03286855
Title: A Randomized Controlled Trial of Bronchodilator Delivery by Vibrating Mesh (VM) Nebuliser Versus Small Volume Nebuliser During an Acute Exacerbation of COPD
Brief Title: Effectiveness of Vibrating Mesh Versus Small Volume Nebuliser in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Collaborators: Aerogen (Industry)
Responsible Party: Principal Investigator, Professor Richard Costello, Consultant Respiratory Physician, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCA NEB
Record Dates: First submitted 2017-09-13; First posted 2017-09-19 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; Copd Exacerbation Acute; COPD Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: prospective feasibility open-label randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vibrating Mesh Group (Experimental): Patient's admitted with an acute exacerbation of COPD and prescribed nebulised combined salbutamol 2.5mg/ipratropium bromide 0.5mg (Combivent) are randomised to receive their treatment via the Aerogen Ultra (CE 0050) vibrating mesh Nebuliser.
  Interventions: Device: Vibrating Mesh Nebuliser
- Standard Hospital Care Group (Active Comparator): Patient's admitted with an acute exacerbation of COPD and prescribed nebulised combined salbutamol 2.5mg/ipratropium bromide 0.5mg (Combivent) are randomised to receive their treatment via the Hudson micromist small volume nebuliser which is the standard of care at our institution.
  Interventions: Device: Standard Hospital Care

INTERVENTIONS:
Device: Vibrating Mesh Nebuliser — The Aerogen Ultra vibrating mesh nebuliser is an approved 13 485 class II medical device (CE marked) nebuliser licenced for the delivery of physician-prescribed medications for inhalation which are approved for use with a general purpose nebuliser. It has been shown in previous laboratory and clinical studies to have superior drug delivery to standard jet nebulisers.
  Other Names: Aerogen Ultra 13 485 class II medical device (CE 0050)
  Arms: Vibrating Mesh Group
Device: Standard Hospital Care — The "standard hospital care" refers to the nebuliser in clinical use currently throughout Beaumont Hospital and used for the administration of nebulised medications. This is the Hudson micromist small volume nebuliser.
  Arms: Standard Hospital Care Group

SUMMARY:
When patients get an attack of COPD, one of the main treatments is regular nebulised medications called bronchodilators. These medications act by opening up the airways allowing patients to breathe easier and to reduce shortness of breath. Newer nebulisers may increase the amount of medication that gets into the lungs compared to the standard nebuliser usually used in hospital. This study is being done to assess whether increasing the amount of medication getting into the lungs using these newer nebulisers will help patients recover from a COPD exacerbation.

DETAILED DESCRIPTION:
COPD is a common chronic respiratory disease. It is characterised by repeated episodes of acute worsening of symptoms of cough, wheeze and breathlessness called exacerbations. Exacerbations result in patients having to present to hospital for treatment. In Ireland more than one-fifth of all inpatient hospital days for the treatment of respiratory complaints are for the treatment of COPD. The administration of bronchodilators (medication to open the airway) is a central component of the treatment of COPD exacerbation. In the hospital setting these are most commonly administered via a nebuliser. The standard of care in our institution is the Hudson micromist small volume nebuliser.

However, previous studies have shown that Vibrating mesh (VM) nebulisers result in greater deposition of medication to the lungs compared to small volume nebulisers. In addition they resulted in greater improvements in lung function and breathlessness.

This study will assess the efficacy of the Aerogen Ultra VM nebuliser in a real-world setting. The VM nebuliser is readily available for use in the clinical setting and is used to administer bronchodilator therapy, within the terms of its CE Mark. This nebuliser is already in routine use in hospitals within the Royal College of Surgeons in Ireland (RCSI) hospital group.

Patients hospitalised with an exacerbation of COPD will be recruited. There will be two study groups. Group 1 (VM Group): will receive bronchodilator (salbutamol 2.5mg/ipratropium 0.5mg) by Vibrating Mesh Nebuliser (Aerogen Ultra) with facemask and Group 2 (Standard Hospital Care): will receive bronchodilator by small volume nebuliser (Hudson Micromist) via facemask as per standard care.

Both groups will receive bronchodilator therapy four times a day which has already been prescribed by their medical team, and in accordance with recommended guidelines for treatment of COPD exacerbations. Patients will use the nebuliser for the duration of hospital stay or a maximum of 7 days. Lung function and breathlessness scores will be recorded. The aim of this study is to demonstrate that better medication delivery by VM nebulizer during an exacerbation of COPD will lead to greater bronchodilation, shorter recovery time and reduced hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Admission with acute exacerbation of COPD within 24 hours of presentation to hospital
* Age >40
* Confirmed COPD diagnosis (FEV1/FVC <0.70 on spirometry)
* Willing to participate in the study and provide informed consent

Exclusion Criteria:

* Admission for reason other than COPD exacerbation e.g. Heart Failure
* Acute confusion as per clinical team
* Allergy or contraindication to combined bronchodilator medication
* Severe respiratory sepsis as evident by temperature >38 degrees and/or lobar pneumonia on Chest Radiograph
* Sustained tachycardia >120bpm
* Patients with very advanced COPD, admitted for palliative or long term care
* Patients re-admitted within 90 days who have already been enrolled in the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Up to 7 days
  Forced spirometry measured at bedside

SECONDARY OUTCOMES:
Change in Borg breathlessness score | Up to 7 days
  Change in patient-reported breathlessness as determined by the Borg breathlessness score
Length of Hospital Stay | Up to 7 days
  Defined as time from randomisation to medical decision to discharge patient
Change in Inspiratory Capacity (IC) | Up to 7 days
  Relaxed spirometry measured at bedside
Rate of re-exacerbation at Day 30 | Up to 30 days
  The number of repeat exacerbations following discharged from hospital. Exacerbation defined as an acute change in respiratory symptoms necessitating administration of antibiotics and/or steroids
Time to re-exacerbation . | Up to 30 days
  The time to first repeat exacerbation following discharge.Exacerbation defined as an acute change in respiratory symptoms necessitating administration of antibiotics and/or steroids
Change in quality of life (QOL): to discharge and to Day 30 | Up to 30 days
  COPD Assessment Test Score
Personal Satisfaction Score | Up to 7 days
  End-user questionnaire
Change in Forced Expiratory Volume in one second (FEV1) | Up to 7 days
  Forced spirometry measured at bedside

CONTACTS AND LOCATIONS:
Overall Officials: Richard W Costello, Principal Investigator — Royal College of Surgeons in Ireland
Locations (1):
- Beaumont Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No